CLINICAL TRIAL: NCT05478629
Title: National Audit of the Safety of Regional Anesthesia in Hospitals of Ukraine
Brief Title: Safety of Regional Anesthesia in Ukraine: the Survey
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Kateryna Bielka, Associate Professor, Bogomolets National Medical University
Other Study IDs: 151
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Regional Anesthesia Morbidity
Keywords: regional anesthesia; LAST; Patient safety
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Questioning through google forms

SUMMARY:
The common using of ultrasound navigation makes an opportunity to develop the regional anesthesia. Regional anesthesia reduces the length of stay in the hospital, reduces the intensity of perioperative pain and decrease opioid using. But systemic toxicity of local anesthetics (LAST) is a significant problem. Prevalence of LAST in Europe range from 0.04 to 1.8 cases per 100 thousand local anesthesia. No similar studies have been provided in Ukraine before, and there are no statistics on the LAST epidemiology. Goal of this survey - evaluation of the prevalence of LAST, the safety of regional anesthesia in Ukraine.

DETAILED DESCRIPTION:
The survey was conducted from October 2021-February 2022 by filling out a standard Google form. The survey design was approved by Bogomolets National Medical University ethical committee (protocol #151 on 25 October 2021). All participants sign the informed consent form before filling out the questionnaire. The link to the survey was published on the Ukrainian Association of Anesthesiologists webpage and Facebook page. The survey link is https://aaukr.org/opytuvannya-shhodo-vypadkiv-toksychnosti-mistsevyh-anestetykiv/.

To conduct the survey, we formed a questionnaire of 14 items. We studied the literature that describes in detail the methods of providing similar surveys [5, 6].

The questionnaire was designed to ensure sufficient collection of data from respondents on demographics, awareness of the LAST guidelines, the availableness of ultrasound navigation, and of preparations of fat emulsions in their departments. Also, we made an accent on the presence of safety protocols, using a check-list of LAST before every regional anesthesia. And we've investigated communication in the hospital if LAST or another critical incident occurs in the OR.

The structure of the questionnaire makes doctors an opportunity to fill it in a short time. We also provided respondents with more descriptive and detailed answers to some questions if they wished. The questionnaire is available in the supplemental material. Multiple options to answer are required to fill, other questions were free to answer. The survey was provided in Ukrainian. Only practicing anesthesiologists, heads of departments, practicing Ph.D. students and professors were invited to take part in the survey.

Statistical analysis. We've imported the results of the survey into Microsoft Excel for continuous analysis. Simple descriptive statistics were used.

ELIGIBILITY:
Inclusion Criteria:

practicing anesthesiologists

Exclusion Criteria:

working not in Ukraine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Practicing anesthesiologists, chiefs of the ICU, teaching assistants
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2023-04-20 (Estimated)

PRIMARY OUTCOMES:
Prevalence of the ultrasound navigation, LAST protocols | 10/01/2021-02/23/2022

CONTACTS AND LOCATIONS:
Locations (1):
- Bogomolets NMU, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The survey link — https://aaukr.org/opytuvannya-shhodo-vypadkiv-toksychnosti-mistsevyh-anestetykiv/